CLINICAL TRIAL: NCT04514939
Title: Elevate to Alleviate - Evidence Based Nursing Study
Brief Title: Elevate to Alleviate Evidence Based Study
Acronym: ETA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.12
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Leg Edema; Venous; Return (Anomaly); Leg Elevation
Keywords: venous returns; lower limbs; leg elevation
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Leg elevation: Patients will lie in their hospital bed with a moderate leg elevation (between 15 and 30 degrees)
  Interventions: Other: Elevation of the legs during bed rest
- Group B- Non Leg elevation: Patients will lie in their hospital bed without leg elevation

INTERVENTIONS:
Other: Elevation of the legs during bed rest — Patients of Group A will will lie in their hospital bed with a moderate leg elevation (between 15 and 30 degrees)
  Groups: Group A - Leg elevation

SUMMARY:
Venous return in the circulatory system of lower limbs results from the interaction of several mechanisms, and reflects the balance between blood inflow and outflow. Blood outflow improves during sleeping because of the lying position especially with leg elevation. In fact, patients with chronic venous disease (CVD) improve leg symptoms in lying position and with leg elevation.

The aim of this study is to evaluate the level of comfort of hospital inpatients, without CVD, if they lie with a moderate leg elevation during hospital stay.

DETAILED DESCRIPTION:
The venous system makes the blood return to the heart with low-pressure and slow-velocity flow, within the venous system. Venous return results from the interaction of diverse mechanisms, such a central pump (respiratory cycle and the heart), a pressure gradient, a peripheral venous muscular pump, and the veins valvular system. Therefore, the venous volume in the lower limb is the result of the interaction between these mechanisms and reflects the balance between blood inflow and outflow. Blood outflow improves during sleeping because of the lying position and, in this position, even more with leg elevation. In fact, it is known patients with chronic venous disease (CVD) improve leg symptoms in lying position and with leg elevation.

The aim of this study is to evaluate the level of comfort of hospital inpatients, without CVD, if they lie with a moderate leg elevation during hospital stay.

Unselected patients with a hospital stay of at least seven days will be recruited and random assigned to two groups of patients: Group A, that will lie in their hospital bed with a moderate leg elevation (between 15 and 30 degrees). Group B, that will lie in their hospital bed without leg elevation.

All patients will undergo echo duplex scanning of vascular system of lower limbs to exclude any vascular disease.

For every patient complete demographic and comorbidity data will be collected. Every single the day, the following parameters will be retrieved for each patient: ankle and calf diameters, heart rate, blood pressure, breath frequency, body temperature, leg heaviness (rating scale 1-10), perceived leg comfort (rating scale 1-10), hours of night sleep (number).

ELIGIBILITY:
Inclusion Criteria:

* Every hospital inpatient with at least 7 hospital stay.

Exclusion Criteria:

* Patients with vascular or osteoarticular leg problems that affect or prevent leg elevation during rest.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Unselected patients with a hospital stay of at least seven days will be recruited and random assigned to two groups of patients of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Ankle and calf diameters measurement | at 6 months
  Every Morning Ankle and calf diameters will be measured in centimeters.
Legs heaviness evaluation | at 6 months
  Every Morning Each patient will comunicate his/her perception of legs heaviness using a rating scale (1-10: 1 is absence of heaviness and 10 is high heaviness)
Perceived leg comfort evaluation | at 6 months
  Every Morning Each patient will comunicate his/her perception of legs heaviness using a rating scale (1-10: 1 is minimum comfort and 10 is maximum comfort)
Hours of night sleep | at 6 months
  Every Morning Each patient will comunicate the number of hours slept

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Ielapi, R.N., Principal Investigator — University of Roma La Sapienza
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liaw MY, Wong MK. [The effects of leg elevation to reduce leg edema resulting from prolonged standing]. Taiwan Yi Xue Hui Za Zhi. 1989 Jun;88(6):630-4, 628. Chinese. PMID 2794965
- [Background] Sugisawa R, Unno N, Saito T, Yamamoto N, Inuzuka K, Tanaka H, Sano M, Katahashi K, Uranaka H, Marumo T, Konno H. Effects of Compression Stockings on Elevation of Leg Lymph Pumping Pressure and Improvement of Quality of Life in Healthy Female Volunteers: A Randomized Controlled Trial. Lymphat Res Biol. 2016 Jun;14(2):95-103. doi: 10.1089/lrb.2015.0045. Epub 2016 Jan 29. PMID 26824795